CLINICAL TRIAL: NCT02193880
Title: Safety of Post-transplant Alpha-beta Depleted T-cell Infusion Following Haploidentical Stem Cell Transplant (Haplo SCT)
Acronym: ABD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayman Saad (Other)
Responsible Party: Sponsor-Investigator, Ayman Saad, Assoc Prof Medicine M.D., University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAB 1397
Record Dates: First submitted 2014-07-14; First posted 2014-07-18 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Hematologic Neoplasms; Graft-Versus-Host Disease
Keywords: stem cell transplant
MeSH Terms: conditions — Hematologic Neoplasms; Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Alpha-beta depleted T-cell infusion (Other): Post-transplant alpha-beta depleted T-cell infusion after post-transplant cyclophosphamide.
  Interventions: Device: Alpha-beta depleted T-cell infusion after post-transplant cyclophosphamide.

INTERVENTIONS:
Device: Alpha-beta depleted T-cell infusion after post-transplant cyclophosphamide. — Post-transplant alpha-beta depleted T-cell infusion after post-transplant cyclophosphamide.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of post-transplant cyclophosphamide and a post-transplant infusion of donor cells, that have been specially processed to remove alpha beta t-cells, in patients undergoing a haploidentical allogeneic stem cell transplant to help reduce the risk of relapse without increasing the risk of graft-versus-host disease.

DETAILED DESCRIPTION:
Transplant patients participating in this clinical trial will receive one of 3 standard pre-transplant chemotherapy preparative regimens as appropriate for their specific disease. They will then receive a standard non-manipulated donor stem cell infusion on transplant day (day 0) followed by cyclophosphamide (days +3 and +4) and an alpha-beta t-cell reduced donor stem cell infusion on day +7.

ELIGIBILITY:
Inclusion Criteria:

* Neoplastic hematological disorder with indication of allogeneic transplant
* No available suitable HLA-matched donor
* Adequate cardiac, pulmonary, renal, and hepatic function
* Karnofsky performance status score greater than or equal to 70%

Exclusion Criteria:

* Medication non-compliance
* No appropriate caregiver identified
* Uncontrolled medical or psychiatric disorder
* Active central nervous system (CNS) neoplastic involvement
* Known allergy to Dimethyl Sulfoxide
* HIV1 or HIV2 positive
* Pregnant or breastfeeding

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-10-09 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Saad, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Medical Center (University of Alabama at Birmingham), Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SJ, Klein J, Haagenson M, Baxter-Lowe LA, Confer DL, Eapen M, Fernandez-Vina M, Flomenberg N, Horowitz M, Hurley CK, Noreen H, Oudshoorn M, Petersdorf E, Setterholm M, Spellman S, Weisdorf D, Williams TM, Anasetti C. High-resolution donor-recipient HLA matching contributes to the success of unrelated donor marrow transplantation. Blood. 2007 Dec 15;110(13):4576-83. doi: 10.1182/blood-2007-06-097386. Epub 2007 Sep 4. PMID 17785583
- [Background] Alshemmari S, Ameen R, Gaziev J. Haploidentical hematopoietic stem-cell transplantation in adults. Bone Marrow Res. 2011;2011:303487. doi: 10.1155/2011/303487. Epub 2011 Jul 13. PMID 22046559
- [Background] Copelan EA. Hematopoietic stem-cell transplantation. N Engl J Med. 2006 Apr 27;354(17):1813-26. doi: 10.1056/NEJMra052638. No abstract available. PMID 16641398
- [Background] Aversa F, Terenzi A, Tabilio A, Falzetti F, Carotti A, Ballanti S, Felicini R, Falcinelli F, Velardi A, Ruggeri L, Aloisi T, Saab JP, Santucci A, Perruccio K, Martelli MP, Mecucci C, Reisner Y, Martelli MF. Full haplotype-mismatched hematopoietic stem-cell transplantation: a phase II study in patients with acute leukemia at high risk of relapse. J Clin Oncol. 2005 May 20;23(15):3447-54. doi: 10.1200/JCO.2005.09.117. Epub 2005 Mar 7. PMID 15753458
- [Background] Gale RP, Horowitz MM. Graft-versus-leukemia in bone marrow transplantation. The Advisory Committee of the International Bone Marrow Transplant Registry. Bone Marrow Transplant. 1990 Jul;6 Suppl 1:94-7. PMID 2390646
- [Background] Horowitz MM, Gale RP, Sondel PM, Goldman JM, Kersey J, Kolb HJ, Rimm AA, Ringden O, Rozman C, Speck B, et al. Graft-versus-leukemia reactions after bone marrow transplantation. Blood. 1990 Feb 1;75(3):555-62. PMID 2297567
- [Background] Ferrara JL, Yanik G. Acute graft versus host disease: pathophysiology, risk factors, and prevention strategies. Clin Adv Hematol Oncol. 2005 May;3(5):415-9, 428. PMID 16167015
- [Background] Oevermann L, Handgretinger R. New strategies for haploidentical transplantation. Pediatr Res. 2012 Apr;71(4 Pt 2):418-26. doi: 10.1038/pr.2011.60. Epub 2012 Jan 25. PMID 22278184
- [Background] Lamb LS Jr, Lopez RD. gammadelta T cells: a new frontier for immunotherapy? Biol Blood Marrow Transplant. 2005 Mar;11(3):161-8. doi: 10.1016/j.bbmt.2004.11.015. PMID 15744234
- [Background] Moretta L, Locatelli F, Pende D, Marcenaro E, Mingari MC, Moretta A. Killer Ig-like receptor-mediated control of natural killer cell alloreactivity in haploidentical hematopoietic stem cell transplantation. Blood. 2011 Jan 20;117(3):764-71. doi: 10.1182/blood-2010-08-264085. Epub 2010 Oct 1. PMID 20889923
- [Background] Palmer JM, Rajasekaran K, Thakar MS, Malarkannan S. Clinical relevance of natural killer cells following hematopoietic stem cell transplantation. J Cancer. 2013;4(1):25-35. doi: 10.7150/jca.5049. Epub 2012 Dec 5. PMID 23386902
- [Background] Lamb LS Jr, Henslee-Downey PJ, Parrish RS, Godder K, Thompson J, Lee C, Gee AP. Increased frequency of TCR gamma delta + T cells in disease-free survivors following T cell-depleted, partially mismatched, related donor bone marrow transplantation for leukemia. J Hematother. 1996 Oct;5(5):503-9. doi: 10.1089/scd.1.1996.5.503. PMID 8938522
- [Background] Lamb LS Jr, Gee AP, Hazlett LJ, Musk P, Parrish RS, O'Hanlon TP, Geier SS, Folk RS, Harris WG, McPherson K, Lee C, Henslee-Downey PJ. Influence of T cell depletion method on circulating gammadelta T cell reconstitution and potential role in the graft-versus-leukemia effect. Cytotherapy. 1999;1(1):7-19. doi: 10.1080/0032472031000141295. PMID 19746645
- [Background] Godder KT, Henslee-Downey PJ, Mehta J, Park BS, Chiang KY, Abhyankar S, Lamb LS. Long term disease-free survival in acute leukemia patients recovering with increased gammadelta T cells after partially mismatched related donor bone marrow transplantation. Bone Marrow Transplant. 2007 Jun;39(12):751-7. doi: 10.1038/sj.bmt.1705650. Epub 2007 Apr 23. PMID 17450185
- [Background] Handgretinger R. New approaches to graft engineering for haploidentical bone marrow transplantation. Semin Oncol. 2012 Dec;39(6):664-73. doi: 10.1053/j.seminoncol.2012.09.007. PMID 23206843
- [Background] Eto M, Mayumi H, Tomita Y, Yoshikai Y, Nishimura Y, Maeda T, Ando T, Nomoto K. Specific destruction of host-reactive mature T cells of donor origin prevents graft-versus-host disease in cyclophosphamide-induced tolerant mice. J Immunol. 1991 Mar 1;146(5):1402-9. PMID 1671578
- [Background] Strauss G, Osen W, Debatin KM. Induction of apoptosis and modulation of activation and effector function in T cells by immunosuppressive drugs. Clin Exp Immunol. 2002 May;128(2):255-66. doi: 10.1046/j.1365-2249.2002.01777.x. PMID 11985515
- [Background] Luznik L, Engstrom LW, Iannone R, Fuchs EJ. Posttransplantation cyclophosphamide facilitates engraftment of major histocompatibility complex-identical allogeneic marrow in mice conditioned with low-dose total body irradiation. Biol Blood Marrow Transplant. 2002;8(3):131-8. doi: 10.1053/bbmt.2002.v8.pm11939602.
- [Background] Luznik L, Jalla S, Engstrom LW, Iannone R, Fuchs EJ. Durable engraftment of major histocompatibility complex-incompatible cells after nonmyeloablative conditioning with fludarabine, low-dose total body irradiation, and posttransplantation cyclophosphamide. Blood. 2001 Dec 1;98(12):3456-64. doi: 10.1182/blood.v98.12.3456. PMID 11719388
- [Background] Mayumi H, Umesue M, Nomoto K. Cyclophosphamide-induced immunological tolerance: an overview. Immunobiology. 1996 Jul;195(2):129-39. doi: 10.1016/S0171-2985(96)80033-7. PMID 8877390
- [Background] Burroughs LM, O'Donnell PV, Sandmaier BM, Storer BE, Luznik L, Symons HJ, Jones RJ, Ambinder RF, Maris MB, Blume KG, Niederwieser DW, Bruno B, Maziarz RT, Pulsipher MA, Petersen FB, Storb R, Fuchs EJ, Maloney DG. Comparison of outcomes of HLA-matched related, unrelated, or HLA-haploidentical related hematopoietic cell transplantation following nonmyeloablative conditioning for relapsed or refractory Hodgkin lymphoma. Biol Blood Marrow Transplant. 2008 Nov;14(11):1279-87. doi: 10.1016/j.bbmt.2008.08.014. PMID 18940683
- [Background] Luznik L, O'Donnell PV, Symons HJ, Chen AR, Leffell MS, Zahurak M, Gooley TA, Piantadosi S, Kaup M, Ambinder RF, Huff CA, Matsui W, Bolanos-Meade J, Borrello I, Powell JD, Harrington E, Warnock S, Flowers M, Brodsky RA, Sandmaier BM, Storb RF, Jones RJ, Fuchs EJ. HLA-haploidentical bone marrow transplantation for hematologic malignancies using nonmyeloablative conditioning and high-dose, posttransplantation cyclophosphamide. Biol Blood Marrow Transplant. 2008 Jun;14(6):641-50. doi: 10.1016/j.bbmt.2008.03.005. PMID 18489989
- [Background] Brunstein CG, Fuchs EJ, Carter SL, Karanes C, Costa LJ, Wu J, Devine SM, Wingard JR, Aljitawi OS, Cutler CS, Jagasia MH, Ballen KK, Eapen M, O'Donnell PV; Blood and Marrow Transplant Clinical Trials Network. Alternative donor transplantation after reduced intensity conditioning: results of parallel phase 2 trials using partially HLA-mismatched related bone marrow or unrelated double umbilical cord blood grafts. Blood. 2011 Jul 14;118(2):282-8. doi: 10.1182/blood-2011-03-344853. Epub 2011 Apr 28. PMID 21527516
- [Background] Alvarnas JC, Brown PA, Aoun P, Ballen KK, Bellam N, Blum W, Boyer MW, Carraway HE, Coccia PF, Coutre SE, Cultrera J, Damon LE, DeAngelo DJ, Douer D, Frangoul H, Frankfurt O, Goorha S, Millenson MM, O'Brien S, Petersdorf SH, Rao AV, Terezakis S, Uy G, Wetzler M, Zelenetz AD, Naganuma M, Gregory KM; National Comprehensive Cancer Network. Acute lymphoblastic leukemia. J Natl Compr Canc Netw. 2012 Jul 1;10(7):858-914. doi: 10.6004/jnccn.2012.0089. PMID 22773801
- [Background] Hoppe RT, Advani RH, Ai WZ, Ambinder RF, Bello CM, Bierman PJ, Blum KA, Dabaja B, Duron Y, Forero A, Gordon LI, Hernandez-Ilizaliturri FJ, Hochberg EP, Maloney DG, Mansur D, Mauch PM, Metzger M, Moore JO, Morgan D, Moskowitz CH, Poppe M, Pro B, Weiss L, Winter JN, Yahalom J; NCCN Hodgkin Lymphoma. Hodgkin lymphoma. J Natl Compr Canc Netw. 2011 Sep 1;9(9):1020-58. doi: 10.6004/jnccn.2011.0086. No abstract available. PMID 21917626
- [Background] Zelenetz AD, Wierda WG, Abramson JS, Advani RH, Andreadis CB, Bartlett N, Bellam N, Byrd JC, Czuczman MS, Fayad LE, Glenn MJ, Gockerman JP, Gordon LI, Harris NL, Hoppe RT, Horwitz SM, Kelsey CR, Kim YH, Krivacic S, LaCasce AS, Nademanee A, Porcu P, Press O, Pro B, Reddy N, Sokol L, Swinnen L, Tsien C, Vose JM, Yahalom J, Zafar N, Dwyer MA, Naganuma M; National Comprehensive Cancer Network. Non-Hodgkin's lymphomas, version 1.2013. J Natl Compr Canc Netw. 2013 Mar 1;11(3):257-72; quiz 273. doi: 10.6004/jnccn.2013.0037. PMID 23486452
- [Background] O'Donnell MR, Tallman MS, Abboud CN, Altman JK, Appelbaum FR, Arber DA, Attar E, Borate U, Coutre SE, Damon LE, Lancet J, Maness LJ, Marcucci G, Martin MG, Millenson MM, Moore JO, Ravandi F, Shami PJ, Smith BD, Stone RM, Strickland SA, Wang ES, Gregory KM, Naganuma M; National Comprehensive Cancer Network. Acute myeloid leukemia, version 2.2013. J Natl Compr Canc Netw. 2013 Sep 1;11(9):1047-55. doi: 10.6004/jnccn.2013.0127. PMID 24029121
- [Background] O'Brien S, Radich JP, Abboud CN, Akhtari M, Altman JK, Berman E, DeAngelo DJ, Deininger M, Devine S, Fathi AT, Gotlib J, Jagasia M, Kropf P, Moore JO, Pallera A, Pinilla-Ibarz J, Reddy VV, Shah NP, Smith BD, Snyder DS, Wetzler M, Gregory K, Sundar H; Ntational comprehensive cancer network. Chronic Myelogenous Leukemia, Version 1.2014. J Natl Compr Canc Netw. 2013 Nov;11(11):1327-40. doi: 10.6004/jnccn.2013.0157. PMID 24225967
- [Background] Greenberg PL, Attar E, Bennett JM, Bloomfield CD, Borate U, De Castro CM, Deeg HJ, Frankfurt O, Gaensler K, Garcia-Manero G, Gore SD, Head D, Komrokji R, Maness LJ, Millenson M, O'Donnell MR, Shami PJ, Stein BL, Stone RM, Thompson JE, Westervelt P, Wheeler B, Shead DA, Naganuma M. Myelodysplastic syndromes: clinical practice guidelines in oncology. J Natl Compr Canc Netw. 2013 Jul;11(7):838-74. doi: 10.6004/jnccn.2013.0104. PMID 23847220
- [Background] Tefferi A. Primary myelofibrosis: 2013 update on diagnosis, risk-stratification, and management. Am J Hematol. 2013 Feb;88(2):141-50. doi: 10.1002/ajh.23384. PMID 23349007
- [Background] Przepiorka D, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995 Jun;15(6):825-8. PMID 7581076
- [Background] Le Tourneau C, Lee JJ, Siu LL. Dose escalation methods in phase I cancer clinical trials. J Natl Cancer Inst. 2009 May 20;101(10):708-20. doi: 10.1093/jnci/djp079. Epub 2009 May 12. PMID 19436029
- [Background] Luznik L, Bolanos-Meade J, Zahurak M, Chen AR, Smith BD, Brodsky R, Huff CA, Borrello I, Matsui W, Powell JD, Kasamon Y, Goodman SN, Hess A, Levitsky HI, Ambinder RF, Jones RJ, Fuchs EJ. High-dose cyclophosphamide as single-agent, short-course prophylaxis of graft-versus-host disease. Blood. 2010 Apr 22;115(16):3224-30. doi: 10.1182/blood-2009-11-251595. Epub 2010 Feb 2. PMID 20124511
- [Background] Kaplan, EL, Meier, P. Nonparametric estimation from incomplete observations. Journal of the American Statistical Association 53(282): 457-481, 1958.
- [Background] Gray, RJ. A class of K-sample tests for comparing the cumulative incidence of a competing risk. The Annals of Statistics, 1141-1154, 1988.
- See also: Click here for more information about the Bone Marrow Transplantation and Cell Therapy Program at the University of Alabama at Birmingham. — http://www.uab.edu/medicine/bonemarrow/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alpha-beta Depleted T-cell Infusion
Started | 7
Completed | 4
Not Completed | 3
Not completed — patients did not collect enough HPC | 3

BASELINE CHARACTERISTICS:
Population: we report data on 4 patients who received the actual therapy. The other 3 patients did not receive the experimental therapy for NOT collecting enough T cells.
Arm/Group | Alpha-beta Depleted T-cell Infusion
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 48 [32 to 55]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: we report data on 4 patients who received the actual therapy. The other 3 patients did not receive the experimental therapy for NOT collecting enough T cells.
  Participants
    Female | 3
    Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experience Acute Haploidentical Alpha Beta Depleted Transplant (aGVHD)
Description: Patients will be monitored for Grade IV aGVHD and organ toxicity. Acute assessment will be done using the modified Keystone (Glucksberg) consensus criteria.
Time Frame: From baseline and before day +100 of transplant.
Population: we report data on 4 patients who received the actual therapy. The other 3 patients did not receive the experimental therapy for NOT collecting enough CD34 HSCT..
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-beta Depleted T-cell Infusion
Number analyzed (Participants) | 4
Participants | 0

2. Primary Outcome: Number of Participants That Experience Chronic Haploidentical Alpha Beta Depleted Transplant (cGVHD)
Description: Patients will be monitored for Grade IV cGVHD and organ toxicity. Chronic assessment will be done using the conventional criteria.
Time Frame: From baseline and before day +100 of transplant.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-beta Depleted T-cell Infusion
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: Baseline through one year.
Arm/Group | Alpha-beta Depleted T-cell Infusion
All-Cause Mortality (participants affected / at risk) | 3/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha-beta Depleted T-cell Infusion (N=4)
Graft Failure (not related to study) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha-beta Depleted T-cell Infusion (N=4)
Infection (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT02193880/Prot_SAP_000.pdf